CLINICAL TRIAL: NCT05521568
Title: Diagnostic Accuracy of Rapid Molecular Tests for Group A Streptococcal Pharyngitis Using Saliva Samples: Prospective Multicenter Study in Primary Care
Brief Title: Diagnostic Accuracy of Rapid Molecular Tests for Group A Streptococcal Pharyngitis Using Saliva Samples
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other); University Hospital, Paris (Other); Groupe Hospitalier Diaconesses Croix Saint-Simon (Other); Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Other Study IDs: PREDISTREP IX
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Streptococcal Pharyngitis
Keywords: sore throat, rapid tests, molecular tests, saliva, sensitivity, specificity
MeSH Terms: conditions — Pharyngitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Double throat swabs will be taken from each participant. One will be used during consultation to perform the rapid antigen detection test. One will be sent to the microbiology laboratory to perform the reference standard test. If the throat swab grows Group A Streptococcus on culture, the strain will be stored at -80°C for 5 years.
  Below we describe 3 Groups to allow a sufficiently detailed description of all tests, but the index test, the reference standard, and the comparator test will be performed on all study participants (i.e., 'single-gate' design).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Index test : Abbott ID NOW STREP A 2
  Interventions: Diagnostic Test: Index test: Abbott ID NOW STREP A 2
- Reference standard test : Composite of culture and PCR-based tests based on a throat swab
  Interventions: Diagnostic Test: Reference standard test: Composite of culture and PCR-based tests based on a throat swab
- Comparator test : Rapid antigen detection test (usual care)
  Interventions: Diagnostic Test: Comparator test: Rapid antigen detection test (usual care)

INTERVENTIONS:
Diagnostic Test: Index test: Abbott ID NOW STREP A 2 — The test under evaluation ('index test') is the rapid molecular test for Group A streptococcus Abbott ID NOW STREP A 2 (performed on saliva samples instead of throat swabs). This test was chosen because of its ease of use and several previous evaluations showing high diagnostic accuracy on throat swabs. The test gives a result after 2 to 6 minutes and will be performed by primary care practitioners participating in the study, in their office, using salivary swabs instead of throat swabs. Investigators will receive one session of specific training prior to the study. Saliva samples will be collected using the cotton swab that comes within the test packages. Index test results will not be used for patient management. Clinicians performing the rapid saliva test will not be blinded to clinical information.
  Groups: Index test : Abbott ID NOW STREP A 2
Diagnostic Test: Reference standard test: Composite of culture and PCR-based tests based on a throat swab — Throat samples will be obtained by use of a double-swab collection-transportation system :
  * Swab #1 will be used to perform the rapid antigen detection test (see below)
  * Swab #2 will be held at ambient temperature and sent within 72 hours to Robert Debre Hospital microbiology laboratory. Throat swabs will be used to perform throat cultures using standard techniques (PMID: 22768060). Throat swabs will also be used to perform a PCR specific for Group A streptococcus (PMID: 23465407). Samples with a positive culture and/or a positive PCR test result will be classified as reference-standard-positives. Samples with a negative culture and a negative PCR will be classified as reference-standard-negatives. Investigators will be blinded to clinical data, including the result of the rapid antigen detection test and the rapid saliva test.
  Groups: Reference standard test : Composite of culture and PCR-based tests based on a throat swab
Diagnostic Test: Comparator test: Rapid antigen detection test (usual care) — As per usual care, all children will undergo a rapid antigen detection test (StreptAtest, Biosynex), using Swab#1 (see above). This rapid antigen detection test is the one used in France and is the only commercial kit that is officially recommended by the National Health Insurance system. It detects Lancefield's Group A antigen, which is specific to Group A Streptococcus. The test will be performed by investigators, during consultation time. Clinicians performing the rapid antigen detection test will not be blinded to clinical information.
  Groups: Comparator test : Rapid antigen detection test (usual care)

SUMMARY:
Observational study evaluating the diagnostic accuracy of rapid point-of-care molecular Group A strep diagnostic tests in saliva as compared to standard culture- and PCR-based techniques for the management of children aged 3-15 years of age presenting with sore throat to primary care.

DETAILED DESCRIPTION:
Group A streptococcus (GAS) is found in 20% to 40% of cases of childhood pharyngitis; the remaining cases are viral. Streptococcal pharyngitis ('strep throat') deserves antibiotics, while these are not indicated in viral cases. Because signs and symptoms of streptococcal and viral cases overlap, most guidelines recommend relying on a diagnostic test to identify Group A streptococcus to select who should receive antibiotics. In most settings, the first-line test to detect Group A Streptococcus is a rapid antigen detection test based on a throat swab, and the reference standard to identify streptococcal cases is throat culture. Recently, new rapid tests were developed. They use molecular techniques, such as rapid PCRs or LAMP, based on throat swabs. We hypothesize that these new molecular tests are sensitive enough to be performed on saliva swabs instead of throat swabs. Collecting saliva is less invasive and could be done by personnel with limited training.

ELIGIBILITY:
Inclusion Criteria:

* children 3-15 years
* seen in primary care (general practitioner or primary care pediatrician)
* with a diagnosis of acute pharyngitis defined as an inflammation of the pharynx and/or tonsils (erythema with or without exudate) or acute sore throat (even if without local signs of pharyngeal inflammation)
* non-opposition of the accompanying parent(s)

Exclusion Criteria:

* children who received antibiotics within 7 days before inclusion
* children already enrolled in the study for the same episode of pharyngitis

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (3 to 15 years) with acute pharyngitis in primary care
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the Abbott ID NOW STREP A 2 rapid molecular test on saliva samples. | Immediatly after the test

SECONDARY OUTCOMES:
Difference in sensitivity between the rapid molecular tests on saliva and the classical rapid antigen detection tests on throat swabs | Immediatly after the test

OTHER OUTCOMES:
Variability in sensitivity and specificity of rapid molecular tests on saliva according to the McIsaac score (modified Centor score) | Immediatly after the test
Time needed to perform the rapid molecular test on saliva and obtain the results | Immediatly after the test
Satisfaction of the physician, the child, and the accompanying parent(s) withe a questionnaire | Through study completion, an average of 1,5 year
Main reasons for not performing rapid tests among primary care practitioners | Through study completion, an average of 1,5 year

CONTACTS AND LOCATIONS:
Locations (1):
- ACTIV, Saint-Maur-des-Fossés, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Touitou R, Bidet P, Dubois C, Partouche H, Bonacorsi S, Jung C, Cohen R, Levy C, Cohen JF. Diagnostic accuracy of a rapid nucleic acid test for group A streptococcal pharyngitis using saliva samples: protocol for a prospective multicenter study in primary care. Diagn Progn Res. 2023 Jul 13;7(1):13. doi: 10.1186/s41512-023-00150-4. PMID 37443047